CLINICAL TRIAL: NCT01712061
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel Group, Multi-center Study To Evaluate The Efficacy And Safety Of Once-daily Administration Of A Chemokine Ccr2/5 Receptor Antagonist (Pf-04634817) In Adults With Type 2 Diabetes And Overt Nephropathy
Brief Title: A Phase 2 Multi-Center Study To Evaluate The Efficacy And Safety Of A Chemokine CCR2/5 Receptor Antagonist In Adults With Type 2 Diabetes And Overt Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1261007; 2012-003332-23 (EudraCT Number)
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Results first posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-09

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic nephropathy; type 2 diabetes; albuminuria; chemokine antagonist
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2; Albuminuria | interventions — PF-04634817

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 PF-04634817 (Active Comparator)
  Interventions: Drug: PF-04634817
- Arm 2 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04634817 — Three or four tablets (50mg) daily for 12 weeks, depending on baseline renal function
  Arms: Arm 1 PF-04634817
Drug: Placebo — Three or four tablets (50mg) daily for 12 weeks, depending on baseline renal function
  Arms: Arm 2 Placebo

SUMMARY:
The study hypothesis under test is that administration of a CCR2/5 antagonist to subjects with type 2 diabetes and overt nephropathy will result in a reduction in urinary albumin, a surrogate for improved glomerular filtration.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes together with stages 2, 3a, 3b or 4 CKD, based on an eGFR of 20-75 mL/min/1.73m2.
* Evidence of persistent, overt albuminuria; defined as a UACR >=300 mg/g (>=33.9 mg/mmol) or UPCR >=390 mg/g (44.1 mg/mmol), or equivalent, for 3 months or longer.
* Stable background therapy of RAAS inhibition (ie, an ACE inhibitor and/or an ARB, which may also include an aldosterone antagonist in double RAAS but not triple RAAS inhibitor therapy) for at least 3 months before screening and to be maintained for the duration of the study.

Exclusion Criteria:

* Subjects with CKD resulting from type 1 diabetes or non-diabetic CKD.
* Subjects who are diagnosed with autosomal dominant polycystic kidney disease (ADPCKD), severe peripheral vascular disease (PVD) or obstructive uropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (142):
- United States (65):
  - Medical Investigations, Inc., Little Rock, Arkansas
  - North America Research Institute, Azusa, California
  - California Institute of Renal Research, Chula Vista, California
  - California Kidney Specialists, Covina, California
  - Diabetes/Lipid Management and Research Center, Huntington Beach, California
  - Tower Nephrology Medical Group, Los Angeles, California
  - Richard S. Cherlin, MD, Los Gatos, California
  - Providence Clinical Research, North Hollywood, California
  - Desert Oasis Healthcare Medical Group, Palm Springs, California
  - Central Coast Nephrology, Salinas, California
  - California Kidney Specialists, San Dimas, California
  - University of Colorado Denver/University of Colorado Hospital, Aurora, Colorado
  - Gulf Coast Endocrine and Diabetes Center, Clearwater, Florida
  - Continental Research Corp., Doral, Florida
  - Premier Research Associate, Inc., Hialeah, Florida
  - Prestige Clinical Research Center, Miami, Florida
  - Elite Clinical Research, Miami, Florida
  - Nephrology Associates of South Miami, Miami, Florida
  - Tellus Clinical Research, Inc., Miami, Florida
  - Ocean Blue Medical Research Center, Inc, Miami Springs, Florida
  - Diabetes Care Center, New Port Richey, Florida
  - Gulf Coast Kidney Center, New Port Richey, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Pines Clinical Research, Inc., Pembroke Pines, Florida
  - Christie Clinic, LLC, Champaign, Illinois
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Crescent City Clinical Research Center, Metairie, Louisiana
  - CTRC, Interim LSU Public Hospital, New Orleans, Louisiana
  - Pharmacy Department, Interim LSU Public Hospital, New Orleans, Louisiana
  - A. Kaldun Nossuli MD Research, Bethesda, Maryland
  - Western New England Renal and Transplant Associates, PC, Springfield, Massachusetts
  - Hurley Medical Center, Flint, Michigan
  - Apex Medical Research, MI, Inc., Flint, Michigan
  - Troy Internal Medicine, PC, Troy, Michigan
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - VA Medical Center, Kansas City, Missouri
  - Creighton Diabetes Center, Omaha, Nebraska
  - Renal Medicine Associates, Albuquerque, New Mexico
  - Winthrop University Hospital, Division of Nephrology and Hypertension, Mineola, New York
  - Winthrop University Hospital, Pharmacy Department, Mineola, New York
  - Northport VA Medical Sciences Center, Northport, New York
  - Mountain Kidney and Hypertension Associates, PA, Asheville, North Carolina
  - East Carolina University Nephrology Research, Greenville, North Carolina
  - Down East Medical Associates, P.A., Morehead City, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - BRAHN-Hypertension and Nephrology, Inc, Providence, Rhode Island
  - South Carolina Nephrology and Hypertension Center, Inc., Orangeburg, South Carolina
  - The Endocrine Clinic, PC, Memphis, Tennessee
  - Nephrology Associates, P.C., Nashville, Tennessee
  - Independent Clinical Research, Greenville, Texas
  - Clinical Trial Network, Houston, Texas
  - Southwest Nephrology Associates, LLP, Houston, Texas
  - Southwest Houston Research LTD, Houston, Texas
  - Southwest Nephrology Associates, LLP, Richmond, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Briggs Clinical Research, LLC, San Antonio, Texas
  - San Antonio Kidney Disease Center Physicians Group, P.L.L.C., San Antonio, Texas
  - Southwest Nephrology Associates, LLP, Sugar Land, Texas
  - Southern Utah Kidney and Hypertension, St. George, Utah
  - Burke Internal Medicine & Research, Burke, Virginia
  - Clinical Research Institute of Northern Virginia, Inc., Burke, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Zablocki Veterans Affairs Medical Center, Milwaukee, Wisconsin
- Argentina (6):
  - Centro de Salud Renal Junin S.R.L., Junín, Buenos Aires
  - Centro de Investigaciones Medicas - Clinica de Fracturas y Ortopedia, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes S.R.L, Quilmes, Buenos Aires
  - Instituto de Cardiologia de Corrientes "Juana Francisca Cabral", Corrientes
  - CETENE S.A. - Centro de Nefrologia y Dialisis, San Miguel de Tucumán
  - Centro de Investigaciones Clinicas del Litoral S.R.L., Santa Fe
- Australia (7):
  - Liverpool Hospital, Liverpool, New South Wales
  - Department of Nephrology, New Lambton, New South Wales
  - Westmead Hospital, Department of Renal Medicine, Westmead, New South Wales
  - Sunshine Coast Hospital & Health Service, Nambour, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (10):
  - Vancouver General Hospital, Vancouver, British Columbia
  - BC Diabetes.ca, Vancouver, British Columbia
  - Co-Medica Research Network Inc., Courtice, Ontario
  - OTT Healthcare Incorporated, Scarborough Village, Ontario
  - Dr. Stephen S. Chow Medicine Professional Corporation, Toronto, Ontario
  - Toronto East General Medical Centre, Toronto, Ontario
  - Centre de Recherche Clinique de Laval, Laval, Quebec
  - Hopital Maisonneuve-Rosemont-Nephrology, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal Centre de recherche, Montreal, Quebec
  - Pro-Recherche, Saint Romuald, Quebec
- Germany (11):
  - Dialysezentrum Elsterland, Herzberg, Brandenburg
  - Studienzentrum Haematologie/Onkologie/Diabetologie, Aschaffenburg
  - Universitatsmedizin Berlin - Charite Campus Mitte, Berlin
  - GWT-TUD GmbH, Dresden
  - Studienzentrum Karlstrasse GmbH, Düsseldorf
  - Profil Institut fuer Stoffwechselforschung GmbH (branch: Diabetes Praxis Essen), Essen
  - Diabetes Schwerpunktpraxis / Zentrum fur Klinische Studien, Falkensee
  - Medizinische Hochschule Hannover, Hanover
  - Nephrologisches Zentrum Hoyerswerda, Hoyerswerda
  - Zentrum Klinische Studien Neuwied, Neuwied
  - Diabetologische Schwerpunktpraxis, Schwabenheim
- Hong Kong (3):
  - Department of Medicine and Therapeutics, Prince of Wales Hospital,, Shatin, New Territories, Hong Kong SAR
  - Department of Medicine and Therapeutics, Shatin, New Territories, Hong Kong SAR
  - Queen Mary Hospital, Hong Kong
- Italy (9):
  - AOU Consorziale Policlinico di Bari, Bari, BA
  - Ospedale Alessandro Manzoni, Lecco, Italy
  - Ospedale Versilia, Lido Camaiore. (Lucca), Lucca
  - *Ospedale Versilia, Lido Di Camaiore (lucca), Lucca
  - Ospedale Versilia, Lido Di Camaiore (lucca), Lucca
  - A.O.U. Policlinico di Modena, Modena, MO
  - Azienda Ospedaliera Ospedali Riuniti di Foggia, Foggia
  - Unita Cardiometabolica e Trials Clinici, Milan
  - Fondazione Salvatore Maugeri Clinica del Lavoro e della Riabilitazione IRCCS, Pavia
- Malaysia (3):
  - Hospital Universiti Sains Malaysia, Kubong Kerian, Kelantan
  - Hospital Taiping, Taiping, Perak
  - Selayang Hospital, Batu Caves, Selangor
- Peru (5):
  - Casa de Diabetes y Nutricion, Lima, Lima Province
  - Consultorio de Endocrinologia - LM Servicios Medicos y Endocrinologicos EIRL, Lima, Lima Province
  - Centro de Investigacion y Atencion Cardiovascular S.A.C. - Clinica Novocardio, Lima
  - Clinica Maison de Sante ¿ Sede este, Lima
  - Clinica Virgen Maria Auxiliadora, Piura
- Poland (8):
  - Krakowskie Centrum Medyczne Sp. z.o.o., Krakow, Lesser Poland Voivodeship
  - Stacja Dializ, Golub-Dobrzyń
  - LANDA Specjalistyczne Gabinety Lekarskie, Krakow
  - SCM Sp. z.o.o, Krakow
  - Klinika Nefrologii, Hipertensjologii i Transplantologii Nerek, Lodz
  - NZOZ TRI-medica, Lodz
  - CSK MSW w Warszawie Klinika Chorob Wewnetrznych Endokrynologii i Diabetologii, Warsaw
  - KO-MED, Central Kliniczne Sp. z.o.o, Zamość
- Puerto Rico (2):
  - Ponce School of Medicine - CAIMED Center, Ponce
  - Medical Sciences Campus University of Puerto Rico, Rio Piedras
- Romania (4):
  - Spital Clinic Municipal "Dr. Gavril Curteanu" Oradea, Oradea, Jud. Bihor
  - Institutul National de Diabet, Nutritie si Boli Metabolice, Bucharest
  - Elit Medical SRL, Diabet Zaharat Nutritie si Boli Metabolice, Ploieşti
  - Spitalul Clinic Judetean de Urgenta Timisoara, Timișoara
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Yonsei University College of Medicine, Severance Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
- Spain (6):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Parc de Salut Mar. Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital Universitario Dr Peset, Valencia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1261007&StudyName=A%20Phase%202%20Multi-Center%20Study%20To%20Evaluate%20The%20Efficacy%20And%20Safety%20Of%20A%20Chemokine%20CCR2/5%20Receptor%20Antagonist%20In%20Adults%20With%20Type%202%20D

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The primary entry criterion for participants was based on presence of macroalbuminuria (urine albumin to creatinine ratio [UACR] greater than or equal to (>=)300 milligrams per gram (mg/g).
Groups:
- PF-04634817 150 mg: Participants with estimated glomerular filtration rate (eGFR) values of 20 to less than (<)30 milliliters/minute (mL/min)/1.73 square meter (m^2) were dosed orally at 150 mg once daily (QD) for 12 weeks.
- PF-04634817 200 mg: Participants with eGFR values of 30 to 75 mL/min/1.73 m^2 were dosed orally at 200 mg QD for 12 weeks.
- Placebo: Participants were dosed orally with matching placebo tablets QD for 12 weeks.
Period: Overall Study
Arm/Group | PF-04634817 150 mg | PF-04634817 200 mg | Placebo
Started | 30 | 140 | 56
Completed | 20 | 114 | 45
Not Completed | 10 | 26 | 11
Not completed — Adverse Event | 4 | 9 | 5
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Did Not Meet Entrance Criteria | 4 | 6 | 3
Not completed — Medication Error Without Associated AE | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 7 | 1
Not completed — Other | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- PF-04634817 200 mg/150 mg: Participants were dosed orally at 150 mg (eGFR 20-<30 mL/min/1.73 m^2) or 200 mg (30-75 mL/min/1.73 m^2) QD for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | PF-04634817 200 mg/150 mg | Placebo | Total
Number analyzed (Participants) | 170 | 56 | 226
Age, Customized [Number; unit: participants]
  Less than (<) 18 years | 0 | 0 | 0
  18-44 years | 3 | 0 | 3
  45-64 years | 78 | 31 | 109
  >=65 years | 89 | 25 | 114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 7 | 43
  Male | 134 | 49 | 183

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction From Baseline in Urinary Albumin to Creatinine Ratio (UACR) at Week 12
Description: The presence of albumin in the urine (macroalbuminuria) is a marker of kidney disease. Albumin and creatinine concentrations were obtained from spot urine samples.
Time Frame: Baseline and Week 12
Population: The Full Analysis Set (FAS) was defined as all participants randomized and who had received at least 1 dose of randomized treatment and had at least 1 post-dose efficacy measurement; n=number of participants analyzed in respective arms for category.
Measure: Mean (95% Confidence Interval); unit: percent (%)
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 159 | 51
percent (%) | 13.27 (5.43) [3.14 to 24.62] | 5.02 (6.87) [-7.90 to 18.70]
Statistical Analysis 1: Comparison: PF-04634817 200 mg/150 mg vs Placebo; Test type: Superiority or Other; ANCOVA; Bayesian ANCOVA with covariates for baseline UACR and systolic blood pressure (SBP); Ratio of geometric mean changes = 0.92, 95% CI 2-sided [0.75 to 1.09]

2. Secondary Outcome: Change From Baseline in UACR at Weeks 4, 8 and 16
Description: as for outcome 1
Time Frame: Baseline, Weeks 4, 8 and 16
Population: The FAS was defined as all participants randomized and who had received at least 1 dose of randomized treatment and had at least 1 post-dose efficacy measurement; n=number of participants analyzed in respective arms for category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/millimolar creatinine (mmolCr)
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 159 | 51
mg/millimolar creatinine (mmolCr)
  Baseline (n=157,50) | 127.41 (96) | 121.80 (88)
  Change From Baseline at Week 4 (n=148,46) | 0.89 (66) | 0.91 (88)
  Change From Baseline at Week 8 (n=134,43) | 0.90 (62) | 0.94 (57)
  Change From Baseline at Week 16 (n=126,37) | 0.93 (72) | 0.92 (56)

3. Secondary Outcome: Change From Baseline in Urinary Protein to Creatinine Ratio (UPCR) at Weeks 4, 8, 12 and 16
Description: The presence of protein in the urine (proteinuria) often implies kidney disease. Protein and creatinine concentrations were obtained from spot urine samples.
Time Frame: Baseline, Weeks 4, 8, 12 and 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/mmolCr
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 159 | 51
mg/mmolCr
  Baseline (n=155,49) | 185.42 (97) | 176.31 (82)
  Change From Baseline at Week 4 (n=143,45) | 0.93 (47) | 0.92 (76)
  Change From Baseline at Week 8 (n=130,42) | 0.92 (50) | 0.94 (46)
  Change From Baseline at Week 12 (n=125,42) | 0.92 (58) | 0.92 (79)
  Change From Baseline at Week 16 (n=125,36) | 0.95 (58) | 0.92 (55)

4. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) Using the Abbreviated Modified Diet in Renal Disease (MDRD) Formula at Weeks 1, 4, 8, 12 and 16
Description: eGFR was calculated using the MDRD equation and normalized to 1.73 m^2 body surface area. Age and corresponding creatinine at each visit (Weeks 1, 4, 8, 12 and 16) were used to calculate GFR
Time Frame: Baseline, Week 1, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 159 | 51
mL/min/1.73m^2
  Baseline (n=159,51) | 41.80 (12.18) | 41.65 (13.46)
  Change From Baseline at Week 1 (n=157,50) | -0.77 (5.80) | -0.35 (5.28)
  Change From Baseline at Week 4 (n=157,51) | -1.07 (5.37) | -1.32 (5.12)
  Change From Baseline at Week 8 (n=147,47) | -1.60 (5.34) | -2.15 (6.83)
  Change From Baseline at Week 12 (n=136,45) | -1.14 (5.70) | -1.03 (5.75)
  Change From Baseline at Week 16 (n=134,44) | -2.14 (6.42) | -1.18 (5.58)

5. Secondary Outcome: Change From Baseline in eGFR Using Cystatin Formula at Weeks 12 and 16
Description: Serum cystatin C may be a more reliable endogenous marker of GFR than serum creatinine. eGFR was calculated using the Cystatin Formula and normalized to 1.73 m^2 body surface area.
Time Frame: Baseline, Week 12, and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 159 | 51
mL/min/1.73m^2
  Baseline (n=159,50) | 45.28 (14.22) | 45.36 (14.94)
  Change From Baseline at Week 12 (n=135,44) | -1.10 (6.30) | -0.70 (5.49)
  Change From Baseline at Week 16 (n=134,43) | -2.27 (6.77) | -0.91 (6.30)

6. Secondary Outcome: Change From Baseline in Serum Creatinine at Weeks 1, 4, 8, 12 and 16
Description: Serum creatinine is an indicator of kidney function. Creatinine is a substance formed from the metabolism of creatine, commonly found in blood, urine, and muscle tissue. It is removed from the blood by the kidneys and excreted in urine. Normal adult blood levels of creatinine=45 to 90 micromoles per liter (mcmol/L) for females, 60 to 110 mcmol/L for males, however normal values are age-dependent. Change from baseline=creatinine level at Week 1, 4, 8, 12 or 16 minus baseline level where higher scores represented decreased kidney function.
Time Frame: Baseline, Week 1, 4, 8, 12 and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 159 | 51
milligrams per deciliter (mg/dL)
  Baseline (n=159,51) | 1.72 (0.51) | 1.77 (0.51)
  Change From Baseline at Week 1 (n=158,50) | 0.05 (0.22) | 0.03 (0.17)
  Change From Baseline at Week 4 (n=157,51) | 0.06 (0.21) | 0.11 (0.30)
  Change From Baseline at Week 8 (n=147,47) | 0.06 (0.21) | 0.09 (0.24)
  Change From Baseline at Week 12 (n=137,45) | 0.05 (0.24) | 0.08 (0.20)
  Change From Baseline at Week 16 (n=134,44) | 0.09 (0.30) | 0.09 (0.29)

7. Secondary Outcome: Change From Baseline in Serum Cystatin C at Weeks 12 and 16
Description: Cystatin C is a protein which is mainly used as a biomarker of kidney function. If kidney function and GFR decline, the blood levels of cystatin C rise.
Time Frame: Baseline, Week 12, and Week 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 159 | 51
mg/dL
  Baseline (n=159,51) | 1.54 (0.43) | 1.52 (0.41)
  Change From Baseline at Week 12 (n=136,45) | 0.03 (0.25) | 0.03 (0.21)
  Change From Baseline at Week 16 (n=134,44) | 0.05 (0.26) | 0.06 (0.25)

8. Secondary Outcome: Change From Baseline in Plasma Glycosylated Hemoglobin (HbA1c) at Weeks 4, 8, 12 and 16
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. As the average amount of plasma glucose increases, the fraction of HbA1c increases in a predictable way.
Time Frame: Baseline, Weeks 4, 8, 12 and 16
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 159 | 51
percent
  Baseline (n=159,51) | 7.51 (1.22) | 7.91 (1.42)
  Change From Baseline at Week 4 (n=157,51) | 0.03 (0.46) | -0.04 (0.46)
  Change From Baseline at Week 8 (n=147,46) | -0.02 (0.64) | -0.08 (0.71)
  Change From Baseline at Week 12 (n=137,44) | -0.01 (0.76) | -0.06 (0.81)
  Change From Baseline at Week 16 (n=133,44) | 0.04 (0.89) | -0.04 (1.13)

9. Secondary Outcome: Summary of Plasma PF-04634817 Pharmacokinetic (PK) Concentrations at Day 1 and Weeks 1, 4, 8 and 12
Time Frame: 1, 2, 4 hours post-dose on Day 1; 2 hours post-dose on Weeks 1, 4, 8 and 12
Population: The PK Concentration Analysis Set is defined as all participants in the FAS for whom a PK sample was obtained and analyzed; n=number of participants analyzed in respective arms for category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-04634817 150 mg | PF-04634817 200 mg
Number analyzed (Participants) | 30 | 140
ng/mL
  Day 1: 1 Hour Post-Dose (n=29,124) | 434.5 (65) | 524.4 (83)
  Day 1: 2 Hours Post-Dose (n=30,139) | 579.3 (37) | 602.9 (52)
  Day 1: 4 Hours Post-Dose (n=29,137) | 497.4 (38) | 547.7 (46)
  Week 1: Pre-Dose (n=28,131) | 294.4 (60) | 231.2 (73)
  Week 1: 2 Hours Post-Dose (n=28,132) | 884.8 (42) | 865.0 (55)
  Week 4: Pre-Dose (n=25,126) | 231.3 (51) | 239.5 (87)
  Week 4: 2 Hours Post-Dose (n=24,122) | 785.8 (45) | 918 (55)
  Week 8: Pre-Dose (n=23,113) | 310.2 (79) | 245.2 (77)
  Week 8: 2 Hours Post-Dose (n=23,114) | 730.0 (70) | 895 (57)
  Week 12 (n=20,113) | 320.1 (75) | 252.3 (84)

10. Other Pre Specified Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Weeks 1, 4, 8, 12 and 16
Time Frame: Baseline, Weeks 1, 4, 8, 12 and 16
Population: The Safety Analysis Set is defined as all participants who receive at least 1 dose of study medication; n=number of participants analyzed in respective arms for category.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 170 | 56
millimeters of mercury (mm Hg)
  Supine SBP: Baseline (n=168,53) | 140.4 (13.96) | 139.9 (13.60)
  Supine SBP:Change From Baseline Week 1 (n=164,53) | -0.8 (12.75) | -1.6 (12.87)
  Supine SBP:Change From Baseline Week 4 (n=154,49) | -0.5 (15.43) | -1.6 (14.19)
  Supine SBP:Change From Baseline Week 8 (n=142,47) | -3.4 (12.94) | -1.1 (13.71)
  Supine SBP:Change From Baseline Week 12 (n=134,45) | -2.0 (13.28) | -1.3 (13.23)
  Supine SBP:Change From Baseline Week 16 (n=138,45) | -2.4 (15.14) | -0.3 (14.41)
  Supine DBP: Baseline (n=168,53) | 75.9 (8.97) | 77.1 (6.88)
  Supine DBP:Change From Baseline Week 1 (n=164,53) | -0.2 (6.94) | -2.7 (7.58)
  Supine DBP:Change From Baseline Week 4 (n=154,49) | 0.1 (8.23) | -1.8 (7.47)
  Supine DBP:Change From Baseline Week 8 (n=142,47) | -1.9 (7.46) | -1.5 (7.05)
  Supine DBP:Change From Baseline Week 12 (n=134,45) | -0.9 (6.88) | -0.2 (6.69)
  Supine DBP:Change From Baseline Week 16 (n=138,45) | -1.7 (7.98) | 0.9 (8.40)

11. Other Pre Specified Outcome: Change From Baseline in Pulse Rate at Weeks 1, 4, 8, 12 and 16
Time Frame: Baseline, Weeks 1, 4, 8, 12 and 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 170 | 56
beats per minute (bpm)
  Baseline (n=168,53) | 68.7 (9.74) | 69.3 (9.30)
  Change From Baseline at Week 1 (n=164,53) | 0.1 (5.86) | -0.7 (5.63)
  Change From Baseline at Week 4 (n=154,49) | 0.3 (6.01) | -1.0 (6.63)
  Change From Baseline at Week 8 (n=142,47) | 0.2 (6.54) | 1.4 (6.77)
  Change From Baseline at Week 12 (n=134,45) | 0.2 (7.03) | 0.5 (7.33)
  Change From Baseline at Week 16 (n=138,45) | 1.4 (8.22) | -0.1 (6.92)

12. Other Pre Specified Outcome: Change From Baseline in Body Weight at Weeks 1, 4, 8, 12 and 16
Time Frame: Baseline, Weeks 1, 4, 8, 12 and 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 170 | 56
kilograms (kg)
  Baseline (n=167,53) | 93.8 (23.97) | 95.1 (25.95)
  Change From Baseline at Week 1 (n=163,53) | 0.0 (1.03) | 0.3 (1.42)
  Change From Baseline at Week 4 (n=153,49) | -0.0 (1.74) | 0.4 (3.29)
  Change From Baseline at Week 8 (n=141,47) | 0.1 (2.45) | 0.7 (2.74)
  Change From Baseline at Week 12 (n=134,45) | 0.3 (2.66) | 0.7 (3.02)
  Change From Baseline at Week 16 (n=137,45) | -0.1 (2.79) | 0.2 (3.37)

13. Other Pre Specified Outcome: Number of Participants With Laboratory Abnormalities Meeting the Criteria for Potential Clinical Concern
Description: The following laboratory parameters were analyzed for abnormalities at any time point mentioned in the timeframe: clinical chemistry (sodium, potassium, chloride, bicarbonate, phosphate, glucose, blood urea nitrogen [BUN], creatinine, albumin, calcium, bilirubin [total, direct, and indirect], gamma-glutamyl transferase [GGT], alanine aminotransferase [ALT], aspartate aminotransferase [AST], lactic dehydrogenase [LDH], alkaline phosphatase, creatine phosphokinase [CPK], uric acid, amylase and lipase); hematology (hemoglobin, hematocrit, red blood cell [RBC] count, white blood cell [WBC] count with differential, and platelet count); FSH (for postmenopausal women who had been amenorrheic for less than 2 years prior to screening).
Time Frame: Baseline up to Week 16 (follow-up visit)
Population: The Safety Analysis Set is defined as all participants who receive at least 1 dose of study medication; number of participants analyzed (N) is number of evaluable participants for this outcome measure.
Measure: Number; unit: participants
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 167 | 53
participants | 154 | 49

14. Other Pre Specified Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings
Description: Criteria for potentially clinically important ECG values were defined as: PR interval >=300 milliseconds (msec) or >=25%/50% increase when baseline is >200 msec and ≥50% increase when baseline is less than or equal to (<=)200 msec; QRS interval >=140 msec or >=50% increase from baseline (IFB); QTc >=450 msec or >=30 msec increase; corrected QT interval using Fridericia's formula (QTcF) >=450 msec or >=30 msec increase.
Time Frame: Baseline, Weeks 1, 4 and 12
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 170 | 56
participants
  Maximum PR Interval >=300 msec (n=164,55) | 3 | 0
  Maximum QRS Complex >=140 msec (n=169,56) | 2 | 1
  Maximum QT Interval >=500 msec (n=169,56) | 0 | 0
  Maximum QTc Interval 450-<480 msec (n=169,56) | 23 | 11
  Maximum QTc Interval 480-<500 msec (n=169,56) | 4 | 1
  Maximum QTc Interval >=500 msec (n=169,56) | 0 | 0
  Maximum QTcF Interval 450-<480 msec (n=169,56) | 11 | 5
  Maximum QTcF Interval 480-<500 msec (n=169,56) | 1 | 1
  Maximum QTcF Interval >=500 msec (n=169,56) | 1 | 0
  PR Interval >=25/50% IFB (n=163,53) | 3 | 0
  QRS Complex >=50% IFB (n=169,55) | 3 | 0
  QTc Interval 30-<60 msec IFB (n=169,55) | 15 | 4
  QTc Interval >=60 msec IFB (n=169,55) | 0 | 0
  QTcF Interval 30-<60 msec IFB (n=169,55) | 8 | 3
  QTcF Interval >=60 msec IFB (n=169,55) | 1 | 0

15. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of treatment and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline up to 28 days after last study drug administration
Population: The Safety Analysis Set is defined as all participants who receive at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 170 | 56
participants
  AEs | 106 | 36
  SAEs | 17 | 5

16. Other Pre Specified Outcome: Number of Participants With Increased Fasting Blood Glucose
Time Frame: Baseline up to Week 16 (follow-up visit)
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | PF-04634817 200 mg/150 mg | Placebo
Number analyzed (Participants) | 167 | 53
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-04634817 150 mg | PF-04634817 200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 6/30 | 11/140 | 5/56
Other Adverse Events (participants affected / at risk) | 11/30 | 40/140 | 15/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04634817 150 mg (N=30) | PF-04634817 200 mg (N=140) | Placebo (N=56)
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 2 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Homicide (Social circumstances) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04634817 150 mg (N=30) | PF-04634817 200 mg (N=140) | Placebo (N=56)
Diarrhoea (Gastrointestinal disorders) | 2 | 12 | 3
Nausea (Gastrointestinal disorders) | 2 | 5 | 2
Oedema peripheral (General disorders) | 3 | 8 | 4
Nasopharyngitis (Infections and infestations) | 2 | 6 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Dizziness (Nervous system disorders) | 2 | 4 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 1
Hypertension (Vascular disorders) | 1 | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.